CLINICAL TRIAL: NCT02774668
Title: A Short Term Evaluation of a Structured Weight Loss Plan in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Principal Investigator, Elizabeth Jane Parks, Professor, Nutrition & Exercise Physiology-MED, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2004733
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome
Keywords: gender; arterial stiffness; blood pressure; weight loss; uric acid
MeSH Terms: conditions — Metabolic Syndrome; Coitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Grab-and-Go" meal plan (Active Comparator): The intervention of this arm is to use a "Grab-and-Go" meal plan. This meal plan provides Atkins shakes and bars for breakfast, lunch, and snacks for 2 weeks. For dinner the subject is given a freshly-prepared meal. Upon finishing the 2-week provided food phase, the subject will consume a self-prepared meal of similar nutrient composition at home for another 2 weeks. For the next four weeks while he/she is still enrolled in the study, he/she will have his/her options for food choices which are not controlled for the study.
  Interventions: Other: "Grab-and-Go" meal plan
- "Jump-Start" meal plan (Active Comparator): The intervention of this arm is to use a "Jump Start" meal plan. This meal plan provides Atkins frozen meals at breakfast, lunch and dinner for 2 weeks and these meals are supplemented with fresh salads and vegetables. Upon finishing the 2-week provided food phase, the subject will consume a self-prepared meal of similar nutrient composition at home for another 2 weeks. For the next four weeks while he/she is still enrolled in the study, he/she will have his/her options for food choices which are not controlled for the study.
  Interventions: Other: "Jump-Start" meal plan

INTERVENTIONS:
Other: "Grab-and-Go" meal plan — The "Grab-and-Go" meal plan will provide Atkins shakes and bars for breakfast, lunch, and snacks. For dinner, the participant will receive a freshly-prepared meal. There will be no difference in terms of calories or nutrient composition between "Grab-and-Go" meal plan versus "Jump-Start" meal plan.
  The amount of weight loss caused by these two meal plans is not expected to differ.
  Arms: "Grab-and-Go" meal plan
Other: "Jump-Start" meal plan — The "Jump-Start" plan will provide Atkins frozen meals at breakfast, lunch and dinner and these meals will be supplemented with fresh salads and vegetables. There will be no difference in terms of calories or nutrient composition between "Grab-and-Go" meal plan versus "Jump-Start" meal plan. The amount of weight loss caused by these two meal plans is not expected to differ.
  Arms: "Jump-Start" meal plan

SUMMARY:
The present study is designed to examine the effect of changes in body weight and related parameters associated with a commercially-available, low-carbohydrate diet plan. A parameter proposed to be studied here is the impact of fructose restriction and weight loss on serum uric acid concentrations and arterial stiffness.

DETAILED DESCRIPTION:
It is well know that consumption of a calorically-restricted diet helps people lose weight. Such a diet with low carbohydrate lowers the serum uric acid concentration which is a factor associated with obesity and also represents a particular metabolic risk in women compared to men. The present weight loss study will determine whether women benefit more than men to short-term weight loss occurring during restriction of simple sugars.

Specifically, this study is designed to cause weight loss acutely through consumption of a diet that is restricted in calorie and simple sugars. Both men and women will be studied and their results compared to determine whether women benefit more with respect to arterial stiffness. Upon finishing the four-week diet intervention, body weight and blood lipids will be assessed two and four weeks later to compare the longer term effect on blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Men and premenopausal women
2. 30-55 years of age
3. Sedentary lifestyle, defined as less than three sessions of activity per week, or sessions less than 20 minutes per occasion, or less than 5000 steps per day
4. Must be able to speak, read, and write English (due to the small sample size and pilot nature of this study)
5. Overweight/obese subjects with BMI 27.0 - 40.0 kg/m2 and any one of the following characteristics of the metabolic syndrome:

A. Serum HDL cholesterol <40 mg/dL (1 mmol/L) in men and <50 mg/dL (1.3 mmol/L) in women B. Blood pressure ≥130/85 mmHg C. Fasting plasma glucose ≥100 mg/dL (5.6 mmol/L) D. Waist circumference in men of >102 cm (40 in) and in women of >88 cm (35 in) E. Serum triglycerides (TG) ≥150 mg/dL (1.7 mmol/L).

Exclusion Criteria:

1. Abnormal thyroid function or known liver disease
2. Diabetes or fasting glucose ≥ 125 mg/dL
3. Use of medications that interfere with protein, carbohydrate or lipid metabolism (e.g., fish oil capsules)
4. Occasional or regular tobacco use
5. History of gout
6. Uncontrolled hypertension
7. Pregnant or peri-menopausal
8. Vegetarian food restrictions (the diets consumed contain some meat, eggs and dairy)
9. Alcohol intake: females > 70 g/wk, males >140 g/wk
10. Moderate or vigorous-intensity physical activity, defined as more than 150 minutes per week of moderate-intensity, or 75 minutes a week of vigorous-intensity aerobic physical activity, or an equivalent combination of both.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Hu, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Syed-Abdul MM, Hu Q, Jacome-Sosa M, Padilla J, Manrique-Acevedo C, Heimowitz C, Parks EJ. Effect of carbohydrate restriction-induced weight loss on aortic pulse wave velocity in overweight men and women. Appl Physiol Nutr Metab. 2018 Dec;43(12):1247-1256. doi: 10.1139/apnm-2018-0113. Epub 2018 May 10. PMID 29746789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the local Columbia, MO area from April 2016 through August 2016
Pre-assignment Details: Subjects underwent screening to assess meeting the eligibility requirements and then were assigned to one of the diet groups. 64 men and women were assessed for eligibility to find the 20 eligible subjects.
Groups:
- "Grab-and-Go" Meal Plan: The intervention of this arm is to use a "Grab-and-Go" meal plan. This meal plan provides Atkins shakes and bars for breakfast, lunch, and snacks for 2 weeks. For dinner the subject is given a freshly-prepared meal. Upon finishing the 2-week provided food phase, the subject will consume a self-prepared meal of similar nutrient composition at home for another 2 weeks. For the next four weeks while he/she is still enrolled in the study, he/she will have his/her options for food choices which are not controlled for the study.
  "Grab-and-Go" meal plan: The "Grab-and-Go" meal plan will provide Atkins shakes and bars for breakfast, lunch, and snacks. For dinner, the participant will receive a freshly-prepared meal. There will be no difference in terms of calories or nutrient composition between "Grab-and-Go" meal plan versus "Jump-Start" meal plan.
  The amount of weight loss caused by these two meal plans is not expected to differ.
Period: Overall Study
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (7.9) | 39.2 (9.0) | 40.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss Between Baseline and 4 Weeks After Completion of Dietary Intervention
Description: For statistical analysis, the body weight is measured at baseline and after 4 weeks after consumption of a calorie-restricted, low-carbohydrate diet.
Time Frame: Change of body weight over 4 weeks of dietary intervention
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan
Number analyzed (Participants) | 10 | 10
kg | 5.5 (1.6) | 5.9 (2.6)

2. Secondary Outcome: Arterial Stiffness Changes Between Baseline and 4 Weeks
Description: Pulse wave velocity, a non-invasive indicator of arterial stiffness will be assessed at the baseline testing and 4 weeks after the start of the dietary intervention.
Time Frame: Arterial stiffness will be measured at baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan
Number analyzed (Participants) | 10 | 10
m/s | -0.4 (0.8) | -0.5 (0.7)

3. Secondary Outcome: Plasma Uric Acid Level Between Baseline and 4 Weeks.
Description: A fasting blood sample will be collected at baseline, 4 weeks after the start of the dietary intervention to measure plasma uric acid level.
Time Frame: Plasma uric acid level will be measured at baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan
Number analyzed (Participants) | 10 | 10
mg/dL | 0.5 (1.4) | 0.04 (1.2)

4. Secondary Outcome: Change in Food Craving Questionnaire (FCI-II-State) at Baseline and 4 Weeks
Description: Food craving questionnaire (FCI-II-State) will be administrated at baseline visit and the end of 4-week after dietary change. Cravings are assessed from 0 (no cravings: "Not at all") to 5 (high cravings:
  "Extremely/Always") for each of the five subscales measures including high-fat foods, sweets, carbohydrates/starches, fast-food fats, and fruits/vegetables. In addition, the scores for each of the subscales were averaged to produce a total cravings measure (also assessed from 0-5).
Time Frame: Questionnaires about food cravings will be administrated at baseline visit and 4 weeks after the start of the meal plan
Population: One subject in the Jump-start arm did not fill out a cravings questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan
Number analyzed (Participants) | 10 | 9
score on a scale | -0.4 (0.6) | -0.3 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the subjects entered baseline testing, during their consumption of the diets, and through the follow-up testing. Because the diets were whole foods, commonly consumed we did not expect many adverse events.
Description: Once a week when the subjects came in to pick up the food, we queried them on constipation, GI effects, and fatigue.
Arm/Group | "Grab-and-Go" Meal Plan | "Jump-Start" Meal Plan
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Limitations are as follows. The loss of weight with low-CHO diet is being assessed over a short period of time. The study has a small sample size and also, it is unknown if these effects would persist with a longer study duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT02774668/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT02774668/ICF_001.pdf